CLINICAL TRIAL: NCT04232592
Title: Clinical Safety Study of Human Embryonic Stem Cell Derived Mesenchymal Cells in the Treatment of Moderate and Severe Intrauterine Adhesions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qi Zhou (Other Government)
Collaborators: Tongji Hospital (Other)
Responsible Party: Sponsor-Investigator, Qi Zhou, Director of Institute of zoology, chinese academy of sciences, and vice president of medical school， University of chinese academy of sciences, Chinese Academy of Sciences
Organization: Chinese Academy of Sciences (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chinese ASZQ-005
Record Dates: First submitted 2019-12-27; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-12

CONDITIONS: Intrauterine Adhesion
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stem cell preparation solution injection group (Experimental): The solution of stem cells preparation will be injected.
  Interventions: Biological: Inject a solution of stem cell preparation
- Injected stem cell group (Experimental): The stem cells will injected.
  Interventions: Biological: Inject stem cells

INTERVENTIONS:
Biological: Inject a solution of stem cell preparation — The control group was injected with a solution of stem cell preparation
  Arms: Stem cell preparation solution injection group
Biological: Inject stem cells — Three dose groups were designed: low dose group, medium dose group and high dose group.
  Arms: Injected stem cell group

SUMMARY:
To observe the clinical safety of intrauterine injection of human embryonic stem cell derived mesenchymal cells in the treatment of moderate and severe intrauterine adhesion, and to preliminarily explore its clinical effectiveness in promoting endometrial regeneration and repair.

DETAILED DESCRIPTION:
In this study, a single-center, controlled, open-label design was used for a dose escalation study.To observe the clinical safety of intrauterine injection of human embryonic stem cell derived mesenchymal cells in the treatment of moderate and severe intrauterine adhesion, and to preliminarily explore its clinical effectiveness in promoting endometrial regeneration and repair.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

* 18 ≤ age ≤38, female;
* According to the 1988 American Fertility Society (AFS) diagnostic criteria, patients with uterine adhesions diagnosed with full civil capacity and with a score of ≥5 were enrolled in the study;
* The patient had one or more of the following clinical symptoms: reduced menstruation or amenorrhea, periodic abdominal pain, secondary infertility, recurrent abortion, premature delivery and other adverse pregnancy outcomes;
* The uterus was smaller than 8 weeks gestation and the uterine cavity depth was less than 12 cm;
* The second to fifth day of menstruation FSH <10mIU/mL, AMH >1.2ng/mL, AFC>6;
* Understand and sign informed consent voluntarily.

Exclusion Criteria:

* Patients with acute pelvic inflammation or endometriosis;
* Having or having a history of malignancy;
* Thrombus, lupus erythematosus and other hormone use contraindications; Allergic to albumin products;
* Patients with uterine malformation, adenomyosis, submucosal uterine fibroids,and uterine fibroids of any site >5cm;
* Patients who were using anticoagulants or who had not recovered normal platelet function 10 days after discontinuation of antiplatelet drugs;
* Previous history of abnormal coagulation function or abnormality before cell transplantation;
* Always has a history of abnormal bleeding (such as abnormal bleeding during tooth extraction), or their immediate family members have hemorrhagic disease,such as hemophilia, bleeding symptoms (e.g., hematemesis, black, serious or recurrent nasal bleeding, coughing up blood, obvious hematuria, gastrointestinal bleeding, or intracranial hemorrhage), or suspected of vascular malformation such as aneurysm by researchers determine influence cell implant operation;
* Alcohol or drug addiction;
* Participated in other interventional clinical trials within 90 days before the informed consent was signed or before the cell transplantation;
* Had used glucocorticoids or immunosuppressive drugs within 12 weeks before signing the informed consent;
* Had used antipsychotic drugs, such as antidepressants and anti-manic drugs, within 12 weeks before signing the informed consent;
* Severe heart failure within 24 weeks before the informed consent;
* Glomerular filtration rate (eGFR) <90ml/min;
* ALT>3 times normal upper limit;
* Concomitant with other serious systemic diseases, such as pulmonary heart disease, severe chronic obstructive pulmonary disease (COPD), etc;
* Patients with severe clinical infection should receive antibiotics within 1 week before signing the informed consent;
* Active infectious diseases, including but not limited to positive human immunodeficiency virus and syphilis antibody;
* The researchers considered poor compliance;
* Other conditions not suitable for participation in this clinical trial.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of different Adverse Events of transplantation of mesenchymal cells from human embryonic stem cells | Within 48 weeks after surgery
  Adverse events (AE), severe adverse events (SAE), and treatment-related adverse events (TEAE) occurred within 48 weeks after surgery.

SECONDARY OUTCOMES:
Normal recovery rate of endometrial thickness | 12 months
  Normal recovery rate of endometrial thickness at 1 and 2 months after surgery will be measured (effective rate = endometrium > 6mm after surgery/all participants ×100%).
recurrence rate of intrauterine adhesions | 12 months
  Recurrence rate of intrauterine adhesions (defined as patients with recurrence of intrauterine adhesions reviewed by hysteroscopy at 1 month/total patients ×100%) will be measured.
Intrauterine adhesions score | 12 months
  Intrauterine adhesions score will be measured according to the American Fertility Society in 1988 diagnostic criteria for intrauterine adhesions.The scores range from 1 to 12. Higher scores mean a worse outcome.
The endometrial biopsies for CD31 | 12 months
  Immunohistochemical results of CD31 during the two endometrial biopsies will be measured.
Menstrual volume change | 12 months
  Menstrual volume change will be assessed according to menstrual blood loss chart.
Clinical pregnancy rate | 12 months
  Clinical pregnancy rate, abortion rate, live birth rate, and sustained pregnancy rate (defined as live pregnancy over 12 weeks) will be assessed.
The endometrial biopsies for estrogen | 12 months
  Estrogen receptor levels during the two endometrial biopsies will be measured.
The endometrial biopsies for Ki67 | 12 months
  Ki67 expression levels during the two endometrial biopsies will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Qi Zhou, Doctor, Principal Investigator — Institute of Zoology, Chinese Academy of Sciences